CLINICAL TRIAL: NCT04297410
Title: 177Lu-PSMA-I&T Radionuclide Neo-Adjuvant Treatment in Patients With Locally Advanced Prostate Cancer Prior to Radical Prostatectomy: Feasibility Trial.
Brief Title: 177Lu-PSMA-I&T Prior to Radical Prostatectomy for Locally Advanced Disease
Acronym: NALuPROST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, golan shay, Director of urologic-oncology service, Principal Investigator, Clinical senior lecturer, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0315-19
Record Dates: First submitted 2019-11-25; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant LuPSMA (Experimental)
  Interventions: Radiation: 177Lu-PSMA-I&T Radionuclide

INTERVENTIONS:
Radiation: 177Lu-PSMA-I&T Radionuclide — Each patient will receive two single doses of 7.4 GBq 177-Lu-PSMA-I&T treatments. The treatments will be given intravenously, 2 weeks apart starting 12 weeks prior to radical prostatectomy.

SUMMARY:
Despite surgical advances, up to 50% of patients with high-risk locally advanced prostate cancer will die from their disease. Drug therapy before surgery has the potential to improve treatment success by lowering tumor volume in the prostate and treating small metastases. PET PSMA is an advanced imaging technique that allows the identification of areas involved by the tumor in the prostate or in the pelvis. This technique is based on the protein PSMA (prostate-specific membrane antigen) which is located on the tumor cells. The presence of PSMA on tumor cells has been recently used for treatment purposes. A chemical element (Lutetium) that binds to PSMA and emits local radiation can destroy tumors cells. This treatment has been used in patients with advanced metastatic disease and showed promising results. The investigators hypothesized that using these particles can improve long term results in patients who undergo surgery for prostate cancer which has not extensively spread. The investigators will assess both the immediate and long-term impact of this novel treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male aged 18 years and older. 2. Patients were diagnosed with high risk localized prostate cancer (cT3/4 and/or Gleason score ≥8 and/or prostate biopsy or PSA ≥ 20 ng/dl) or loco-regional prostate cancer (pelvic lymphadenopathy of ≥2 cm on axial imaging).

  3. High PSMA expression was confirmed. PET PSMA with tracer uptake greater than normal liver (maximal standardized uptake value ≥1.5 of liver). In addition, no PET FDG positive sites without high PSMA expression.

  4. Patients should have an Eastern Cooperative Oncology Group (ECOG) performance status score5 of 1 or lower and life expectancy of > 10 years.

Exclusion Criteria:

* 1. Clinically significant impaired bone marrow defined by platelet count lower than 150×103/µl, white blood cells count lower than 4×103/µl, hemoglobin concentration lower than 12mg/dl.

  2. Impaired liver function defined by albumin concentration lower than 3.5 gr/dl.

  3. Impaired kidney function defined by glomerular filtration rate (GFR) lower than 40 mL/min.

  4. Recent radiotherapy (within two months) 5. Concomitant usage of nephrotoxic drugs 6. Evidence of distant metastatic disease (distal lymphadenopathy, visceral or bone metastases).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Surgical safety | 2 years
  Surgical safety will be assessed according to the rate of intra- and post operative complications graded according to the clavien dindo classification.
Early oncological outcomes | 2 years
  Early oncological outcomes will be assessed according to the final surgical histology (e.g. stage , grade) and postoperative PSA

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Beilinson hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No